CLINICAL TRIAL: NCT03050541
Title: The Effects of 3,4-methylenedioxy-N-methylamphetamine (MDMA) on Encoding, Consolidation, and Retrieval of Emotional and Social Memories
Brief Title: Effects of MDMA on Emotional and Social Memories
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 14-1485
Record Dates: First submitted 2014-12-18; First posted 2017-02-13 (Actual); Results first posted 2018-06-29 (Actual); Last update posted 2018-06-29 (Actual); Status verified 2018-05

CONDITIONS: Healthy
Keywords: MDMA; adult
MeSH Terms: interventions — N-Methyl-3,4-methylenedioxyamphetamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- MDMA at Memory Encoding (Experimental): 20 healthy adult volunteers will be randomly assigned to the encoding group (MDMA at Encoding). This group will receive capsules before viewing the study materials, and at retrieval two days later, but they will receive MDMA only in the capsule appropriate to their condition, and the next session capsule will contain placebo.
  Interventions: Drug: MDMA; Drug: Placebo
- MDMA at Memory Retrieval (Experimental): 20 healthy adult volunteers will be randomly assigned to the retrevial group (MDMA at Retrevial). This group will receive placebo before viewing the study materials, and MDMA at retrieval two days later..
  Interventions: Drug: MDMA; Drug: Placebo
- Placebo at both sessions (Placebo Comparator): 20 healthy adult volunteers will be randomly assigned to the placebo group (no drug at either session). This group will receive only placebo during study, session before viewing the study materials, and at retrieval two days later.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MDMA — This is a between subjects, double-blind, placebo controlled design. We are administering oral MDMA to healthy volunteers to measure its effects on the encoding, consolidation, and retrieval stages of memory.
  Arms: MDMA at Memory Encoding; MDMA at Memory Retrieval
Drug: Placebo

SUMMARY:
The purpose of this study is to examine the effects of MDMA on encoding and retrieval of emotional and social memories in healthy young adults. The study will explore the effects on memory retrieval when the drug is administered 1) before encoding, and 2) before retrieval.

DETAILED DESCRIPTION:
Here, we aim to investigate the effects of MDMA (1 mg/kg) on the encoding and retrieval of positive, negative, social, and neutral memories. The study will use a between subjects design with three groups (N = 20 per group). Two of the groups will be randomly assigned to receive MDMA before one of the two stages of memory: Encoding (ENC) or Retrieval (RET). The third group will receive placebo only (PLC). All three groups will receive capsules before viewing the study materials, and at retrieval two days later, but they will receive MDMA only in the capsule appropriate to their condition, and other capsules will contain placebo.

Participants will participate in two sessions: a viewing session during which they will view emotional and neutral stimuli, followed 48 hours later by a retrieval session, during which there will be a surprise memory test with two components (verbally cued recollection and picture recognition). On all sessions subjects will also complete mood questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Normal healthy males and females, aged 18-40 years.

Exclusion Criteria:

1. any current medical condition requiring medication or abnormal electrocardiogram
2. current or past medical condition considered to be a contraindication for the study conditions
3. any current Axis I psychiatric disorder (APA, 1994) including Substance Use Disorder, or Anxiety Disorder or Major Depression in the past year, any history of psychosis
4. less than high school education
5. lack of fluency in English
6. night shift work
7. pregnancy, lactation, or plans to become pregnant
8. use of hormonal contraception

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2014-12; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harriet de Wit, PhD, Principal Investigator — University of Chicago; David Gallo, PhD, Principal Investigator — University of Chicago

RESULTS

PARTICIPANT FLOW:
Groups:
- MDMA at Memory Encoding: 20 healthy adult volunteers will be randomly assigned to the encoding group (MDMA at Encoding). This group will receive capsules before viewing the study materials, and at retrieval two days later, but they will receive MDMA only in the capsule appropriate to their condition, and the next session capsule will contain placebo.
  Oral MDMA: This is a between subjects, double-blind, placebo controlled design. We are administering oral MDMA to healthy volunteers to measure its effects on the encoding, consolidation, and retrieval stages of memory.
  Placebo
- MDMA at Memory Retrievial: 20 healthy adult volunteers will be randomly assigned to the retrevial group (MDMA at Retrevial). This group will receive placebo before viewing the study materials, and MDMA at retrieval two days later..
  Oral MDMA: This is a between subjects, double-blind, placebo controlled design. We are administering oral MDMA to healthy volunteers to measure its effects on the encoding, consolidation, and retrieval stages of memory.
  Placebo
- Placebo at Both Sessions: 20 healthy adult volunteers will be randomly assigned to the placebo group (no drug at either session). This group will receive only placebo during study, session before viewing the study materials, and at retrieval two days later.
  Placebo
Period: Overall Study
Arm/Group | MDMA at Memory Encoding | MDMA at Memory Retrievial | Placebo at Both Sessions
Started | 28 | 28 | 28
Completed | 20 | 20 | 20
Not Completed | 8 | 8 | 8

BASELINE CHARACTERISTICS:
Groups:
- Healthy Adult Volunteers-Oral MDMA at Memory Encoding: 20 healthy adult volunteers will be randomly assigned to the encoding group (MDMA at Encoding). This group will receive capsules before viewing the study materials, and at retrieval two days later, but they will receive MDMA only in the capsule appropriate to their condition, and the next session capsule will contain placebo.
  Oral MDMA: This is a between subjects, double-blind, placebo controlled design. We are administering oral MDMA to healthy volunteers to measure its effects on the encoding, consolidation, and retrieval stages of memory.
  Placebo
- Healthy Adult Volunteers-Oral MDMA at Memory Retrievial: 20 healthy adult volunteers will be randomly assigned to the retrevial group (MDMA at Retrevial). This group will receive placebo before viewing the study materials, and MDMA at retrieval two days later..
  Oral MDMA: This is a between subjects, double-blind, placebo controlled design. We are administering oral MDMA to healthy volunteers to measure its effects on the encoding, consolidation, and retrieval stages of memory.
  Placebo
- Healthy Adult Volunteers-Placebo at Both Sessions: 20 healthy adult volunteers will be randomly assigned to the placebo group (no drug at either session). This group will receive only placebo during study, session before viewing the study materials, and at retrieval two days later.
  Placebo
- Total: Total of all reporting groups
Arm/Group | Healthy Adult Volunteers-Oral MDMA at Memory Encoding | Healthy Adult Volunteers-Oral MDMA at Memory Retrievial | Healthy Adult Volunteers-Placebo at Both Sessions | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 20 | 60
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 10 | 30
  Male | 10 | 10 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: Probability of Accurately Recalling Visual Stimuli
Description: During encoding, participants were presented with labels that were sometimes followed by pictures. During the first memory test, participant were presented again with all of the labels and asked, "Did you see this picture?" Hit and false alarm rates were then calculated, and memory accuracy was measured by hits minus false alarms.
Time Frame: 90 minutes into Session 2
Measure: Mean (Standard Deviation); unit: probability
Arm/Group | Healthy Adult Volunteers-Oral MDMA at Memory Encoding | Healthy Adult Volunteers-Oral MDMA at Memory Retrievial | Healthy Adult Volunteers-Placebo at Both Sessions
Number analyzed (Participants) | 20 | 20 | 20
probability | .52 (.11) | .50 (.16) | .54 (.17)

2. Secondary Outcome: Probability of Accurately Recognizing Visual Stimuli
Description: After the cued recollection task, all of the pictures were presented to participants (i.e., the ones that they had seen, as well as the ones that were not seen). Participants were then asked, "Did you see this picture?" Hit and false alarm rates were calculated, and memory accuracy was measured as hits minus false alarms.
Time Frame: 90 minutes into Session 2
Measure: Mean (Standard Deviation); unit: probability
Arm/Group | Healthy Adult Volunteers-Oral MDMA at Memory Encoding | Healthy Adult Volunteers-Oral MDMA at Memory Retrievial | Healthy Adult Volunteers-Placebo at Both Sessions
Number analyzed (Participants) | 20 | 20 | 20
probability | .82 (.09) | .81 (.15) | .84 (.11)

ADVERSE EVENTS:
Arm/Group | Healthy Adult Volunteers-Oral MDMA at Memory Encoding | Healthy Adult Volunteers-Oral MDMA at Memory Retrievial | Healthy Adult Volunteers-Placebo at Both Sessions
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/0
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes